CLINICAL TRIAL: NCT00851331
Title: Genetic Basis of Idiopathic Focal Epilepsies With Cognitif Deficits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Other Study IDs: 3391
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Epilepsy
Keywords: Benign childhood epilepsy
MeSH Terms: conditions — Epilepsy

INTERVENTIONS:
Genetic: genome analyzes (genetic defects and pathophysiological mechanisms )

SUMMARY:
Epilepsy is a frequent neurological disease in childhood, characterized by recurrent seizures and sometimes with major effects on social, behavioral and cognitive development. Childhood focal epilepsies particularly are age-related diseases mainly occurring during developmental critical period. A complex interplay between brain development and maturation processes and susceptibility genes may contribute to the development of various childhood epileptic syndromes associated with language and cognitive deficits. Indeed, the Landau-Kleffner syndrome (LKS), the continuous spike-and-waves during sleep syndrome (CSWS), and the benign childhood epilepsy with centrotemporal spikes (BCECTS) or benign rolandic epilepsy, are different syndromes that are considered as part of a single continuous spectrum of disorders. While genetic component in those three syndromes remains elusive, novel and high throughput genome analyzes could bring interesting insights into the possible genetic defects and pathophysiological mechanisms underlying and linking the various disorders associating epilepsy with speech and cognitive impairments.

ELIGIBILITY:
Inclusion Criteria:

* iodiopathic focal epilepsy with cognitif deficit

Exclusion Criteria:

* medical history of status epilepticus

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Edouard HIRSCH, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (4):
- France (4):
  - Hôpital Femme Mère Enfant - Hospices Civils de Lyon, Service Epilepsie, Sommeil et Exploration fonctionnelle neurologique pédiatrique, Bron, 69500
  - American Memorial Hospital, CHU de Reims, Unité de Neurologie Pédiatrique - Service Pédiatrie A, Reims
  - Clinique neurologique, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital de Hautepierre, Service de pédiatrie 1, Strasbourg